CLINICAL TRIAL: NCT00783692
Title: A Phase 3, Randomized, Placebo-Controlled, Blinded, Multicenter Study of the Induction and Maintenance of Clinical Response and Remission by Vedolizumab (MLN0002) in Patients With Moderate to Severe Crohn's Disease
Brief Title: Study of Vedolizumab (MLN0002) in Patients With Moderate to Severe Crohn's Disease
Acronym: GEMINI II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: C13007; 2008-002783-33 (EudraCT Number); U1111-1157-7675 (Registry Identifier: WHO); CTRI/2009/091/000135 (Registry Identifier: CTRI); NMRR-08-1047-2202 (Registry Identifier: NMRR); 09/H1102/65 (Registry Identifier: NRES); NL25208.096.08 (Registry Identifier: CCMO); C13007CTIL (Other: Israel MoH)
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; LDP-02

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vedolizumab (Experimental): In the Induction Phase participants received vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2 (Days 1 and 15).
  In the Maintenance Phase, participants who demonstrated a clinical response at Week 6 according to protocol-specified criteria were randomized in a 1:1:1 ratio to double-blind treatment with vedolizumab administered every 4 weeks, vedolizumab administered every 8 weeks, or placebo for up to Week 50. Participants who did not demonstrate response at Week 6 of the Induction Phase continued treatment with vedolizumab, administered every 4 weeks during the Maintenance Phase.
  Interventions: Drug: vedolizumab
- Placebo (Placebo Comparator): In the Induction Phase participants received placebo intravenous infusion at Week 0 and Week 2 (Days 1 and 15). Participants continued to receive placebo during the Maintenance Phase, regardless of treatment response during Induction.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: vedolizumab — Vedolizumab for intravenous infusion
  Other Names: Entyvio; MLN0002; MLN02; LDP-02
  Arms: Vedolizumab
Other: Placebo — Placebo intravenous infusion
  Arms: Placebo

SUMMARY:
The primary purpose of this study was to determine the effect of vedolizumab induction treatment on clinical response and remission at 6 weeks and to determine the effect of vedolizumab maintenance treatment on clinical remission at 52 weeks.

DETAILED DESCRIPTION:
Study C13007 comprised 2 randomized, double-blind, placebo-controlled studies conducted under 1 protocol which, operationally, consisted of 2 phases.

* The Induction Phase, designed to establish the efficacy and safety of vedolizumab for the induction of clinical response and clinical remission, and
* The Maintenance Phase, designed to establish the efficacy and safety of vedolizumab for the maintenance of clinical response and clinical remission.

The 6-week Induction Phase contained 2 cohorts of participants: Cohort 1 participants were randomized and treated with double-blind study drug, and Cohort 2 participants were treated with open-label vedolizumab. The second cohort was enrolled to ensure that the sample size of Induction Phase responders randomized into the Maintenance Study provided sufficient power for the Maintenance Study primary efficacy analysis. These participants did not contribute to the efficacy analyses performed for the Induction Study. Participants in both cohorts were assessed for treatment response at Week 6.

In the Maintenance Phase vedolizumab-treated participants from both Cohort 1 and Cohort 2 who demonstrated a clinical response were randomized in a 1:1:1 ratio to double-blind treatment with vedolizumab administered every 4 weeks (Q4W), vedolizumab administered every 8 weeks (Q8W), or placebo. Vedolizumab-treated participants who did not demonstrate response at Week 6 continued treatment with open-label vedolizumab, administered Q4W. Participants treated with double-blind placebo in the Induction Phase continued on double-blind placebo during the Maintenance Phase, regardless of treatment response during induction. The Maintenance Phase began at Week 6 and concluded with Week 52 assessments.

After the Week 52 assessments, participants may have been eligible to enroll in Study C13008 (NCT00790933; Long-term Safety Study) to receive open-label vedolizumab treatment. Participants who withdrew early (prior to Week 52) due to sustained nonresponse, disease worsening, or the need for rescue medications may have been eligible to enroll in Study C13008. Participants who did not enroll into Study C13008 were to complete a final on-study safety assessment at Week 66 (or Final Safety visit 16 weeks after the last dose) in the Maintenance Phase of Study C13007.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 80
2. Diagnosis of moderately to severely active Crohn's disease (CD)
3. CD involvement of the ileum and/or colon
4. Demonstrated, over the previous 5 year period, an inadequate response to, loss of response to, or intolerance of at least 1 of the following agents, within protocol-specified parameters:

   1. Immunomodulators
   2. Tumor necrosis factor-alpha (TNFα) antagonists
   3. Corticosteroids
5. May be receiving a therapeutic dose of conventional therapies for irritable bowel disease (IBD) defined by the protocol

Exclusion Criteria

1. Evidence of abdominal abscess at the initial screening visit, other than a minimum of 10 aphthous ulcerations involving a minimum of 10 contiguous cm of intestine
2. Extensive colonic resection, subtotal or total colectomy
3. History of >3 small bowel resections or diagnosis of short bowel syndrome
4. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine
5. Have received non permitted IBD therapies within either 30 or 60 days, depending on the medication, as stated in the protocol
6. Chronic hepatitis B or C infection
7. Active or latent tuberculosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 2008-12; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (114):
- United States (110):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Apex Clinical Trials, Birmingham, Alabama
  - Gastrointestinal Bioscience, Los Angeles, California
  - Paramount Medical Specialty, Montebello, California
  - Capital Gastroenterology Consultants Medical Group, Sacramento, California
  - Clinical Applications Laboratories Inc., San Diego, California
  - Desta Digestive Disease Medical Center, San Diego, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Rocky Mountain Clinical Research, LLC, Golden, Colorado
  - Gastroenterology of the Rockies, Lafayette, Colorado
  - Arapahoe Gastroenterology Associates P.C., Littleton, Colorado
  - South Denver Gastroenterology, Lone Tree, Colorado
  - Lynn Institute of Pueblo, Pueblo, Colorado
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Gastroenterology Center of Connecticut, P.C., Hamden, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Jacksonville, Florida
  - East Coast Institute for Research, Jacksonville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - Osler Clinical Research, Melbourne, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - United Medical Research Institute, New Smyrna Beach, Florida
  - Compass Research LLC, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - West Wind'r Research & Development, LLC, Tampa, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Digestive Research Associates, Newnan, Georgia
  - St. Joseph's/Candler Health System, Savannah, Georgia
  - DLW Research System, Snellville, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Carle Clinic Association P.C., Urbana, Illinois
  - Indianapolis Gastroenterology & Hepatology, Inc.- ARC, Indianapolis, Indiana
  - Digestive & Liver Consultants, Clive, Iowa
  - Iowa Digestive Disease Center, Clive, Iowa
  - University Of Kansas, Kansas City, Kansas
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Gastroenterology Associates, Baton Rouge, Louisiana
  - Metropolitan Gastroenterology Group, P.C., Chevy Chase, Maryland
  - Shah Associates, Prince Frederick, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - The Center for Clinical Studies, Dearborn, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Digestive Health Specialists, Tupelo, Mississippi
  - Truman Medical Center, Kansas City, Missouri
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Washington University, St Louis, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Affiliates in Gastroenterology PA, Morristown, New Jersey
  - University of Medicine and Dentistry of New Jersey-NJMS, New Brunswick, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - Hepatobiliary Associates of New York, Bayside, New York
  - Digestive Health Physician, Cheektowaga, New York
  - Long Island Clinical Research Associates, Great Neck, New York
  - Long Island Gastroenterology Group, P.C., Merrick, New York
  - New York Presbyterian Hospital, New York, New York
  - Present Chapman Marion Steinlauf MD PC, New York, New York
  - Kim, Chung MD (Private Practice), Pittsford, New York
  - University of Rochester, Rochester, New York
  - Long Island Digestive Disease Consultants, Setauket, New York
  - SUNY Stony Brook University Medical Center, Stony Brook, New York
  - Syracuse Gastroenterological Associates, Syracuse, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroentology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Northwest Piedmont Clinical Research, Inc., Elkin, North Carolina
  - Burke Research Associates, Morganton, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Dayton Science Institute, Dayton, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - The Oregon Clinic-West Hills Gastroenterology, Portland, Oregon
  - University of Pittsburgh Medical Center - Cancer Centers, Pittsburgh, Pennsylvania
  - Medical University Of SC CAR, Charleston, South Carolina
  - Consultants in Gastroenterology, Columbia, South Carolina
  - Gastroenterology Center of the MidSouth, PC, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Gastroenterology, PA, Austin, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Gastroenterology Consultants, Houston, Texas
  - Jacon Medical Research Associates, Houston, Texas
  - Digestive Health Center, Pasadena, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Stone Oak Research Foundation, San Antonio, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Granite Peaks Gastroenterology, Sandy City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Digestive and Liver Disease Specialist Ltd., Norfolk, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
  - Puget Sound Medical Research, Edmonds, Washington
  - Pharmaseek, LLC, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - GI Research, Edmonton, Alberta
  - Zeidler Ledcor Center-Univerisity of Alberta, Edmonton, Alberta
  - Royal University Hospital, Saskatoon, Saskatchewan
- Pharmaseek, LLC, Ponce, Puerto Rico

REFERENCES:
- [Derived] Wyant T, Yang L, Rosario M. Comparison of the ELISA and ECL Assay for Vedolizumab Anti-drug Antibodies: Assessing the Impact on Pharmacokinetics and Safety Outcomes of the Phase 3 GEMINI Trials. AAPS J. 2020 Nov 16;23(1):3. doi: 10.1208/s12248-020-00518-0. PMID 33200296
- [Derived] Okamoto H, Dirks NL, Rosario M, Hori T, Hibi T. Population pharmacokinetics of vedolizumab in Asian and non-Asian patients with ulcerative colitis and Crohn's disease. Intest Res. 2021 Jan;19(1):95-105. doi: 10.5217/ir.2019.09167. Epub 2020 Jul 10. PMID 32635680
- [Derived] Sands BE, Van Assche G, Tudor D, Akhundova-Unadkat G, Curtis RI, Tan T. Vedolizumab in Combination With Corticosteroids for Induction Therapy in Crohn's Disease: A Post Hoc Analysis of GEMINI 2 and 3. Inflamm Bowel Dis. 2019 Jul 17;25(8):1375-1382. doi: 10.1093/ibd/izy384. PMID 30615117
- [Derived] Feagan BG, Sandborn WJ, Colombel JF, Byrne SO, Khalid JM, Kempf C, Geransar P, Bhayat F, Rubin DT. Incidence of Arthritis/Arthralgia in Inflammatory Bowel Disease with Long-term Vedolizumab Treatment: Post Hoc Analyses of the GEMINI Trials. J Crohns Colitis. 2019 Jan 1;13(1):50-57. doi: 10.1093/ecco-jcc/jjy125. PMID 30203005
- [Derived] Feagan BG, Lasch K, Lissoos T, Cao C, Wojtowicz AM, Khalid JM, Colombel JF. Rapid Response to Vedolizumab Therapy in Biologic-Naive Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2019 Jan;17(1):130-138.e7. doi: 10.1016/j.cgh.2018.05.026. Epub 2018 May 29. PMID 29857145
- [Derived] Feagan BG, Schwartz D, Danese S, Rubin DT, Lissoos TW, Xu J, Lasch K. Efficacy of Vedolizumab in Fistulising Crohn's Disease: Exploratory Analyses of Data from GEMINI 2. J Crohns Colitis. 2018 Apr 27;12(5):621-626. doi: 10.1093/ecco-jcc/jjy019. PMID 29471381
- [Derived] Colombel JF, Sands BE, Rutgeerts P, Sandborn W, Danese S, D'Haens G, Panaccione R, Loftus EV Jr, Sankoh S, Fox I, Parikh A, Milch C, Abhyankar B, Feagan BG. The safety of vedolizumab for ulcerative colitis and Crohn's disease. Gut. 2017 May;66(5):839-851. doi: 10.1136/gutjnl-2015-311079. Epub 2016 Feb 18. PMID 26893500
- [Derived] Rosario M, Dirks NL, Gastonguay MR, Fasanmade AA, Wyant T, Parikh A, Sandborn WJ, Feagan BG, Reinisch W, Fox I. Population pharmacokinetics-pharmacodynamics of vedolizumab in patients with ulcerative colitis and Crohn's disease. Aliment Pharmacol Ther. 2015 Jul;42(2):188-202. doi: 10.1111/apt.13243. Epub 2015 May 20. PMID 25996351
- [Derived] Sandborn WJ, Feagan BG, Rutgeerts P, Hanauer S, Colombel JF, Sands BE, Lukas M, Fedorak RN, Lee S, Bressler B, Fox I, Rosario M, Sankoh S, Xu J, Stephens K, Milch C, Parikh A; GEMINI 2 Study Group. Vedolizumab as induction and maintenance therapy for Crohn's disease. N Engl J Med. 2013 Aug 22;369(8):711-21. doi: 10.1056/NEJMoa1215739. PMID 23964933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 285 investigative sites worldwide from 23 December 2008 to 08 May 2012. The Induction Phase contained 2 cohorts. The eligibility criteria for both cohorts were identical. The purpose of Cohort 2 was to provide enough responders to power the Maintenance Phase primary efficacy analysis.
Pre-assignment Details: In Cohort 1, eligible patients who met entry criteria were randomized to treatment with double-blind vedolizumab 300 mg or placebo in a 3:2 ratio. All Cohort 2 patients were treated with open-label vedolizumab. In the Maintenance Phase participants were assigned to treatment groups based on their Induction Phase treatment and response to therapy.
Groups:
- Placebo: In the Induction Phase participants in Cohort 1 were randomized to receive double-blind placebo intravenous infusions at Week 0 and Week 2. Participants continued to receive placebo every 4 weeks from Week 6 through Week 50 during the Maintenance Phase, regardless of treatment response during induction.
- Induction Phase: DB Vedolizumab: In the Induction Phase participants in Cohort 1 were randomized to receive double-blind (DB) vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2.
- Induction Phase: OL Vedolizumab: In the Induction Phase participants in Cohort 2 received open-label (OL) vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2.
- Maintenance Phase: Placebo: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with placebo every 4 weeks up to Week 50 during the Maintenance Phase.
- Maintenance Phase: Vedolizumab Q8W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with vedolizumab 300 mg every 8 weeks (Q8W) at Weeks 6, 14, 22, 30, 38, and 46, and, to maintain blinding, placebo infusions at Weeks 10, 18, 26, 34, 42, and 50.
- Maintenance Phase: Vedolizumab Q4W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with vedolizumab 300 mg every 4 weeks (Q4W) from Week 6 to Week 50.
- Maintenance Phase: Non-Responders: Participants who received vedolizumab during the Induction Phase who did not demonstrate a clinical response at Week 6 received open-label treatment with vedolizumab 300 mg every 4 weeks from Week 6 to Week 50.
Period: Induction Phase
Arm/Group | Placebo | Induction Phase: DB Vedolizumab | Induction Phase: OL Vedolizumab | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab Q8W | Maintenance Phase: Vedolizumab Q4W | Maintenance Phase: Non-Responders
Started | 148 | 220 | 748 | 0 | 0 | 0 | 0
Treated | 148 | 220 | 747 | 0 | 0 | 0 | 0
Completed | 137 | 199 | 674 | 0 | 0 | 0 | 0
Not Completed | 11 | 21 | 74 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 9 | 24 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 3 | 28 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 9 | 16 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Placebo | Induction Phase: DB Vedolizumab | Induction Phase: OL Vedolizumab | Maintenance Phase: Placebo | Maintenance Phase: Vedolizumab Q8W | Maintenance Phase: Vedolizumab Q4W | Maintenance Phase: Non-Responders
Started | 137 | 0 | 0 | 153 | 154 | 154 | 412
Completed | 42 | 0 | 0 | 64 | 73 | 82 | 163
Not Completed | 95 | 0 | 0 | 89 | 81 | 72 | 249
Not completed — Adverse Event | 7 | 0 | 0 | 15 | 12 | 9 | 38
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 2 | 3 | 4
Not completed — Lack of Efficacy | 79 | 0 | 0 | 64 | 58 | 48 | 177
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 7 | 6 | 9 | 24
Not completed — Lost to Follow-up | 2 | 0 | 0 | 1 | 3 | 2 | 5
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Induction Phase Safety Population, defined as all participants, in both Cohort 1 and Cohort 2, who received any amount of study drug in the Induction Phase (Weeks 0 to 6), according to the actual study drug received.
Groups:
- Placebo: In the Induction Phase participants in Cohort 1 were randomized to receive double-blind placebo intravenous infusions at Week 0 and Week 2.
- Total: Total of all reporting groups
Arm/Group | Placebo | Induction Phase: DB Vedolizumab | Induction Phase: OL Vedolizumab | Total
Number analyzed (Participants) | 148 | 220 | 747 | 1115
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (13.16) | 36.3 (11.57) | 35.6 (12.01) | 36.1 (12.12)
Age, Customized [Number; unit: participants]
  < 35 years | 67 | 111 | 404 | 582
  ≥ 35 years | 81 | 109 | 343 | 533
Age, Customized [Number; unit: participants]
  < 65 years | 142 | 218 | 732 | 1092
  ≥ 65 years | 6 | 2 | 15 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 115 | 401 | 595
  Male | 69 | 105 | 346 | 520
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 19 | 26
  Not Hispanic or Latino | 139 | 214 | 712 | 1065
  Unknown or Not Reported | 4 | 4 | 16 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 124 | 182 | 689 | 995
  Black | 3 | 3 | 17 | 23
  Asian | 19 | 35 | 35 | 89
  Other | 2 | 0 | 6 | 8
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 10 | 30 | 45
  Austria | 4 | 3 | 7 | 14
  Belgium | 12 | 17 | 41 | 70
  Bulgaria | 5 | 7 | 2 | 14
  Canada | 22 | 12 | 103 | 137
  Czech Republic | 11 | 16 | 53 | 80
  Denmark | 0 | 2 | 8 | 10
  Estonia | 1 | 2 | 3 | 6
  France | 4 | 3 | 37 | 44
  Germany | 0 | 1 | 49 | 50
  Greece | 0 | 0 | 2 | 2
  Hong Kong | 2 | 0 | 0 | 2
  Hungary | 9 | 17 | 47 | 73
  Iceland | 0 | 0 | 4 | 4
  India | 10 | 19 | 5 | 34
  Ireland | 0 | 0 | 2 | 2
  Israel | 2 | 4 | 12 | 18
  Italy | 1 | 0 | 13 | 14
  Korea, Republic of | 3 | 12 | 11 | 26
  Latvia | 0 | 2 | 0 | 2
  Malaysia | 1 | 3 | 5 | 9
  Netherlands | 0 | 0 | 7 | 7
  New Zealand | 4 | 5 | 3 | 12
  Norway | 0 | 0 | 13 | 13
  Poland | 7 | 6 | 14 | 27
  Romania | 0 | 1 | 4 | 5
  Russian Federation | 4 | 9 | 15 | 28
  Serbia | 0 | 0 | 3 | 3
  Singapore | 1 | 0 | 0 | 1
  Slovakia | 3 | 5 | 10 | 18
  South Africa | 3 | 3 | 14 | 20
  Spain | 1 | 0 | 6 | 7
  Sweden | 0 | 1 | 8 | 9
  Switzerland | 0 | 1 | 9 | 10
  Taiwan | 0 | 0 | 3 | 3
  Turkey | 2 | 3 | 1 | 6
  Ukraine | 3 | 4 | 9 | 16
  United Kingdom | 0 | 0 | 6 | 6
  United States | 28 | 52 | 188 | 268
Body Weight [Mean (Standard Deviation); unit: kg] | 68.7 (18.90) | 67.1 (19.07) | 70.8 (19.56) | 69.8 (19.42)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (5.77) | 23.1 (5.62) | 24.2 (6.02) | 23.9 (5.93)
Duration of Crohn's Disease (CD) [Mean (Standard Deviation); unit: years] | 8.2 (7.80) | 9.2 (8.18) | 9.2 (7.63) | 9.0 (7.77)
Duration of Crohn's Disease - Categorical [Number; unit: participants]
  < 1 year | 12 | 12 | 45 | 69
  ≥ 1 to < 3 years | 27 | 48 | 126 | 201
  ≥ 3 to < 7 years | 45 | 49 | 191 | 285
  ≥ 7 years | 64 | 111 | 385 | 560
Baseline Disease Activity - Crohn's Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: units on a scale] — Number of participants for whom baseline CDAI scores were available were 147, 219, and 743, respectively.
  The CDAI is a numerical calculation derived from the sum of products from a list of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to ~600 points with lower scores indicating disease remission and higher scores indicating disease worsening.
  units on a scale | 324.6 (78.08) | 327.3 (70.67) | 322.2 (67.17) | 323.6 (69.37)
Baseline Disease Activity - Categorical [Number; unit: participants]
  CDAI ≤ 330 | 81 | 119 | 418 | 618
  CDAI > 330 | 66 | 100 | 325 | 491
  Missing | 1 | 1 | 4 | 6
Baseline C-reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] — Baseline CRP data was only available for 147 participants in the placebo arm.
  mg/L | 23.6 (27.85) | 24.1 (27.23) | 20.4 (27.40) | 21.5 (27.45)
Baseline CRP - Categorical [Number; unit: participants]
  ≤ 2.87 mg/L | 20 | 37 | 130 | 187
  > 2.87 to ≤ 5 mg/L | 14 | 25 | 75 | 114
  > 5 to ≤ 10 mg/L | 28 | 38 | 160 | 226
  > 10 mg/L | 85 | 120 | 382 | 587
  Missing | 1 | 0 | 0 | 1
Baseline Fecal Calprotectin [Mean (Standard Deviation); unit: μg/g] — Number of participants for whom baseline fecal calprotectin data were available were 142, 210, and 719, respectively.
  μg/g | 1421.2 (2076.11) | 1839.9 (2624.92) | 1050.1 (1558.93) | 1254.2 (1908.82)
Baseline Fecal Calprotectin - Categorical [Number; unit: participants]
  ≤ 250 μg/g | 34 | 51 | 201 | 286
  > 250 to ≤ 500 μg/g | 27 | 25 | 112 | 164
  > 500 μg/g | 81 | 134 | 406 | 621
  Missing | 6 | 10 | 28 | 44
Disease Localization [Number; unit: participants]
  Ileum only | 21 | 37 | 123 | 181
  Colon only | 43 | 62 | 211 | 316
  Ileocolonic (both ileum and colon) | 84 | 121 | 413 | 618
History of Prior Surgery for Crohn's Disease [Number; unit: participants]
  Yes | 54 | 98 | 314 | 466
  No | 94 | 122 | 433 | 649
History of Fistulizing Disease [Number; unit: participants]
  Yes | 56 | 90 | 264 | 410
  No | 92 | 130 | 483 | 705
Draining Fistula at Baseline [Number; unit: participants]
  Yes | 23 | 38 | 104 | 165
  All Closed | 2 | 1 | 8 | 11
  No | 123 | 181 | 635 | 939
Smoking Status [Number; unit: participants]
  Current smoker | 34 | 54 | 210 | 298
  Nonsmoker (never smoked) | 85 | 120 | 351 | 556
  Former smoker | 29 | 46 | 185 | 260
  Missing | 0 | 0 | 1 | 1
Baseline Extraintestinal Manifestations [Number; unit: participants]
  Yes | 107 | 133 | 456 | 696
  No | 41 | 87 | 291 | 419
History of Extraintestinal Manifestations [Number; unit: participants]
  Yes | 123 | 177 | 619 | 919
  No | 25 | 43 | 128 | 196

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Percentage of Participants Achieving Clinical Remission at Week 6
Description: Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) score ≤ 150 points.
  The CDAI is used to quantify the symptoms of patients with Crohn's disease and consists of eight factors, each summed after adjustment with a weighting factor. The components of the CDAI are:
  * Number of liquid or soft stools each day for 7 days;
  * Abdominal pain (graded from 0-3 on severity) each day for 7 days;
  * General well-being, subjectively assessed from 0 (well) to 4 (terrible) each day for 7 days;
  * Presence of complications;
  * Taking Lomotil or opiates for diarrhea;
  * Presence of an abdominal mass (0 as none, 2 as questionable, 5 as definite);
  * Hematocrit of < 0.47 in men and < 0.42 in women;
  * Percentage deviation from standard weight.
  The total score ranges from 0 to approximately 600 and with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving clinical remission.
Time Frame: Week 6
Population: Induction Study Intention to Treat (ITT) Population, which consisted of all randomized patients in Cohort 1 who received any amount of blinded study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants in Cohort 1 received double-blind placebo intravenous infusions at Week 0 and Week 2 in the Induction Phase.
- DB Vedolizumab: Participants in Cohort 1 received double-blind vedolizumab 300 mg, administered by intravenous infusion at Week 0 and Week 2 in the Induction Phase.
Arm/Group | Placebo | DB Vedolizumab
Number analyzed (Participants) | 148 | 220
percentage of participants | 6.8 [2.7 to 10.8] | 14.5 [9.9 to 19.2]
Statistical Analysis 1: Comparison: Placebo vs DB Vedolizumab; The Hochberg method was applied to control the overall Type I error rate at a 5% significance level for the multiple comparisons of the primary endpoints. If both p-values were ≤ 0.05, both primary endpoints were to be declared significant. If 1 of the p-values for the primary endpoints was > 0.05, the other p-value was to be tested at the 0.025 level and declared significant only if the p-value was ≤ 0.025. If neither primary was declared significant, no further testing was to be conducted; Test type: Superiority or Other; p = 0.0206, Cochran-Mantel-Haenszel — P-value is based on the Cochran-Mantel-Haenszel (CMH) chi-square test, with stratification according to: 1) concomitant use of oral corticosteroids (yes/no); 2) previous exposure to TNFα antagonists and/or concomitant immunomodulator use (yes/no); Risk Difference (RD) = 7.8, 95% CI 2-sided [1.2 to 14.3] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo

2. Primary Outcome: Induction Phase: Percentage of Participants With Enhanced Clinical Response at Week 6
Description: Enhanced clinical response is defined as a CDAI score at least 100 points lower than Baseline. The CDAI is used to quantify the symptoms of patients with Crohn's disease and consists of eight factors, each summed after adjustment with a weighting factor. The components of the CDAI are:
  * Number of liquid or soft stools each day for 7 days;
  * Abdominal pain (graded from 0-3 on severity) each day for 7 days;
  * General well-being, subjectively assessed from 0 (well) to 4 (terrible) each day for 7 days;
  * Presence of complications;
  * Taking Lomotil or opiates for diarrhea;
  * Presence of an abdominal mass (0 as none, 2 as questionable, 5 as definite);
  * Hematocrit of < 0.47 in men and < 0.42 in women;
  * Percentage deviation from standard weight.
  The total score ranges from 0 to 600 with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving enhanced clinical response.
Time Frame: Baseline and Week 6
Population: Induction Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | DB Vedolizumab
Number analyzed (Participants) | 148 | 220
percentage of participants | 25.7 [18.6 to 32.7] | 31.4 [25.2 to 37.5]
Statistical Analysis 1: Comparison: Placebo vs DB Vedolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2322, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = 5.7, 95% CI 2-sided [-3.6 to 15.0] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo

3. Primary Outcome: Maintenance Phase: Percentage of Participants Achieving Clinical Remission at Week 52
Description: Clinical remission is defined as a CDAI score ≤ 150. The CDAI is used to quantify the symptoms of patients with Crohn's disease and consists of eight factors, each summed after adjustment with a weighting factor. The components of the CDAI are:
  * Number of liquid or soft stools each day for 7 days;
  * Abdominal pain (graded from 0-3 on severity) each day for 7 days;
  * General well-being, subjectively assessed from 0 (well) to 4 (terrible) each day for 7 days;
  * Presence of complications;
  * Taking Lomotil or opiates for diarrhea;
  * Presence of an abdominal mass (0 as none, 2 as questionable, 5 as definite);
  * Hematocrit of < 0.47 in men and < 0.42 in women;
  * Percentage deviation from standard weight.
  The total score ranges from 0 to 600 with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving clinical remission.
Time Frame: Week 52
Population: Maintenance Study ITT Population, defined as all randomized participants who received vedolizumab during the Induction Phase and met the protocol definition of clinical response at Week 6, as assessed by the investigator, were randomized, and received any amount of double-blind study drug in the Maintenance Phase.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with placebo every 4 weeks up to Week 50 during the Maintenance Phase.
- Vedolizumab Q8W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with vedolizumab 300 mg every 8 weeks (Q8W) from Week 6 to Week 50.
- Vedolizumab Q4W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were then randomized to receive double-blind treatment with vedolizumab 300 mg every 4 weeks (Q4W) from Week 6 to Week 50.
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 153 | 154 | 154
percentage of participants | 21.6 [15.1 to 28.1] | 39.0 [31.3 to 46.7] | 36.4 [28.8 to 44.0]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; The Hochberg method was applied to control the overall Type I error rate at a 5% significance level. If both p-values were ≤ 0.05, both dose regimens were to be declared significant. If 1 of the p-values for the 2 dose comparisons was > 0.05, the other p-value was to be tested at the 0.025 level and declared significant only if the p-value was ≤ 0.025. If neither dose was declared significant for the primary endpoint, no further testing was to be conducted; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel — CMH chi-square test, stratified by: 1) concomitant use of oral corticosteroids (yes/no); 2) previous exposure to TNFα antagonists and/or concomitant immunomodulator use (yes/no); 3) enrollment in Cohort 1 or Cohort 2 in the Induction Phase; Risk Difference (RD) = 17.4, 95% CI 2-sided [7.3 to 27.5] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0042, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 14.7, 95% CI 2-sided [4.6 to 24.7] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo

4. Secondary Outcome: Induction Phase: Change From Baseline in C-Reactive Protein (CRP) Levels at Week 6
Description: C-reactive protein (CRP) is a protein found in the blood, the levels of which rise in response to inflammation. Normal concentration in healthy human serum is usually lower than 10 mg/L, slightly increasing with age. Higher levels indicate mild inflammation (10-40 mg/L) and active inflammation (40-200 mg/L).
Time Frame: Baseline and Week 6
Population: Induction Study ITT Population; last observation carried forward (LOCF) imputation was used. Baseline CRP was missing for one participant in the placebo group.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Placebo | DB Vedolizumab
Number analyzed (Participants) | 147 | 220
mg/L | -0.5 [-27.6 to 12.1] | -0.9 [-20.6 to 10.3]
Statistical Analysis 1: Comparison: Placebo vs DB Vedolizumab; If at least 1 of the primary endpoints was significant, the sequential Hochberg procedure was to be used to test the secondary endpoint for significance at the 0.05% level; Test type: Superiority or Other; p = 0.9288, Wilcoxon (Mann-Whitney) — Wilcoxon Rank Sum test on the CRP change from baseline values (two-sided)

5. Secondary Outcome: Maintenance Phase: Percentage of Participants With Enhanced Clinical Response at Week 52
Description: Enhanced clinical response is defined as a CDAI score at least 100 points lower than the Baseline value. The CDAI is used to quantify the symptoms of patients with Crohn's disease and consists of eight factors, each summed after adjustment with a weighting factor. The components of the CDAI are:
  * Number of liquid or soft stools each day for 7 days;
  * Abdominal pain (graded from 0-3 on severity) each day for 7 days;
  * General well-being, subjectively assessed from 0 (well) to 4 (terrible) each day for 7 days;
  * Presence of complications;
  * Taking Lomotil or opiates for diarrhea;
  * Presence of an abdominal mass (0 as none, 2 as questionable, 5 as definite);
  * Hematocrit of < 0.47 in men and < 0.42 in women;
  * Percentage deviation from standard weight.
  The total score ranges from 0 to 600 with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving enhanced clinical response.
Time Frame: Baseline and Week 52
Population: Maintenance Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Vedolizumab Q8W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were randomized to receive double-blind treatment with vedolizumab 300 mg every 8 weeks (Q8W) from Week 6 to Week 50.
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 153 | 154 | 154
percentage of participants | 30.1 [22.8 to 37.3] | 43.5 [35.7 to 51.3] | 45.5 [37.6 to 53.3]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; To maintain the overall Type I error rate at 5% in the multiple-dose comparisons in each key secondary endpoint, the Hochberg method was used. To further maintain the overall Type I error rate at 5%, the key secondary assessments were performed sequentially. The first key secondary endpoint was tested only if 1 or both of the primary comparisons were significant and the next key secondary endpoint was to be tested only if the previous key secondary endpoint was significant for at least 1 dose; Test type: Superiority or Other; p = 0.0132, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 13.4, 95% CI 2-sided [2.8 to 24.0] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0053, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 15.3, 95% CI 2-sided [4.6 to 26.0] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo

6. Secondary Outcome: Maintenance Phase: Percentage of Participants in Corticosteroid-free Clinical Remission at Week 52
Description: Participants using oral corticosteroids at Baseline, who discontinued corticosteroids and were in clinical remission (CDAI score ≤ 150) at Week 52 achieved corticosteroid-free clinical remission. The CDAI quantifies the symptoms of patients with Crohn's disease and consists of eight factors, summed after adjustment with a weighting factor. The total score ranges from 0 to 600 with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving corticosteroid-free clinical remission.
Time Frame: Week 52
Population: Maintenance Study ITT Population, participants who were on corticosteroids at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were randomized to receive double-blind treatment with placebo every 4 weeks up to Week 50 during the Maintenance Phase.
- Vedolizumab Q4W: Participants who received vedolizumab during the Induction Phase and demonstrated a clinical response at Week 6 were randomized to receive double-blind treatment with vedolizumab 300 mg every 4 weeks (Q4W) from Week 6 to Week 50.
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 82 | 82 | 80
percentage of participants | 15.9 [7.9 to 23.8] | 31.7 [21.6 to 41.8] | 28.8 [18.8 to 38.7]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0154, Cochran-Mantel-Haenszel — P-value is based on the CMH chi-square test, with stratification according to: 1) previous exposure to TNFα antagonists and/or concomitant immunomodulator use (yes/no); 2) enrollment in Cohort 1 or Cohort 2 in the Induction Phase; Risk Difference (RD) = 15.9, 95% CI 2-sided [3.0 to 28.7] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0450, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Risk Difference (RD) = 12.9, 95% CI 2-sided [0.3 to 25.5] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo

7. Secondary Outcome: Maintenance Phase: Percentage of Participants With Durable Clinical Remission
Description: Durable clinical remission is defined as CDAI score ≤ 150 points at 80% or more of study visits during the Maintenance Phase, including the Week 52 visit (11 of 13 study visits). The CDAI quantifies the symptoms of patients with Crohn's disease and consists of eight factors, summed after adjustment with a weighting factor. The total score ranges from 0 to 600 with higher scores indicating greater disease activity.
  All participants who prematurely discontinued for any reason were considered as not achieving durable clinical remission
Time Frame: Assessed every 4 weeks from Week 6 to Week 50, and at Week 52
Population: Maintenance Study ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Vedolizumab Q8W | Vedolizumab Q4W
Number analyzed (Participants) | 153 | 154 | 154
percentage of participants | 14.4 [8.8 to 19.9] | 21.4 [14.9 to 27.9] | 16.2 [10.4 to 22.1]
Statistical Analysis 1: Comparison: Placebo vs Vedolizumab Q8W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1036, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 7.2, 95% CI 2-sided [-1.5 to 16.0] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo
Statistical Analysis 2: Comparison: Placebo vs Vedolizumab Q4W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.6413, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Risk Difference (RD) = 2.0, 95% CI 2-sided [-6.3 to 10.2] — Risk Difference = adjusted (for stratification factors) percent vedolizumab - adjusted percent placebo

ADVERSE EVENTS:
Time Frame: From the start of the Induction Phase until a final on-study safety assessment at Week 66 (or Final Safety visit 16 weeks after the last dose).
Groups:
- Placebo: Participants who received double-blind placebo intravenous infusions in the Induction Phase and continued to receive placebo during the Maintenance Phase.
- VDZ/PBO: Participants who received vedolizumab during the Induction Phase and were then randomized to receive placebo during the Maintenance Phase.
- VDZ/VDZ: Participants who received vedolizumab during the Induction Phase and continued to receive vedolizumab during the Maintenance Phase. This includes participants who had a clinical response at Week 6 and were randomized to vedolizumab every 4 weeks or every 8 weeks in the Maintenance Phase, participants who did not achieve a clinical response at Week 6 and continued to receive vedolizumab every 4 weeks for the duration of the study, and participants who withdrew during the Induction phase.
Arm/Group | Placebo | VDZ/PBO | VDZ/VDZ
Serious Adverse Events (participants affected / at risk) | 23/148 | 23/153 | 199/814
Other Adverse Events (participants affected / at risk) | 96/148 | 96/153 | 476/814
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=148) | VDZ/PBO (N=153) | VDZ/VDZ (N=814)
Crohn's disease (Gastrointestinal disorders) | 13 | 8 | 99
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 6
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Ileal stenosis (Gastrointestinal disorders) | 0 | 2 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1 | 2
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Colon dysplasia (Gastrointestinal disorders) | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 16
Abdominal abscess (Infections and infestations) | 0 | 2 | 5
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Appendicitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 2
Device related infection (Infections and infestations) | 0 | 1 | 1
Abscess intestinal (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Latent tuberculosis (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Ureter abscess (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 2
Oedema peripheral (General disorders) | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 4
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cyclic neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Somatoform disorder (Psychiatric disorders) | 0 | 0 | 1
Stress (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 2
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Clostridium test positive (Investigations) | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — This event occurred while the participant was receiving placebo.
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=148) | VDZ/PBO (N=153) | VDZ/VDZ (N=814)
Nausea (Gastrointestinal disorders) | 12 | 18 | 88
Crohn's disease (Gastrointestinal disorders) | 28 | 23 | 84
Abdominal pain (Gastrointestinal disorders) | 21 | 18 | 79
Vomiting (Gastrointestinal disorders) | 10 | 13 | 48
Diarrhoea (Gastrointestinal disorders) | 5 | 12 | 31
Abdominal pain upper (Gastrointestinal disorders) | 4 | 8 | 20
Nasopharyngitis (Infections and infestations) | 10 | 14 | 100
Upper respiratory tract infection (Infections and infestations) | 11 | 5 | 54
Pyrexia (General disorders) | 17 | 22 | 102
Fatigue (General disorders) | 5 | 9 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 21 | 110
Arthritis (Musculoskeletal and connective tissue disorders) | 9 | 2 | 23
Headache (Nervous system disorders) | 19 | 28 | 97
Anaemia (Blood and lymphatic system disorders) | 9 | 5 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.